CLINICAL TRIAL: NCT00172523
Title: Metabolic Disorders in Polycystic Ovarian Syndrome
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9361701094
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2005-09-15 (Estimated); Status verified 2004-10

CONDITIONS: Polycystic Ovary Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
The purpose of this study is to elucidate the significance of adipocytokine in women with PCOS among adiposity, hyperandrogenism and insulin resistance.

DETAILED DESCRIPTION:
Polycystic ovary syndrome (PCOS) is the most common endocrinopathy in women of reproductive age with a probable prevalence of 5% to 10%. PCOS is characterized by chronic anovulation, menstrual irregularities, evidence of hyperandrogenism (either clinical, manifested as hirsutism, acne, male pattern balding, or biochemical, manifested by elevated serum adrenal and/or ovarian androgen concentration). Fifty percent of all patients with PCOS are obese, and the presence of obesity affects the clinical manifestations of PCOS. The underlying pathogenic mechanisms appear to involve insulin resistance and hyperinsulinemia, the magnitude of which is greater in obese than in non-obese women with PCOS.

ELIGIBILITY:
Inclusion Criteria:

* 1. Oligomenorrhea ( less than 6 times spontaneous MC per year) or Amenorrhea. 2. Hyperandrogenism (either clinical or biochemistry. 3. PCO by ultrasound. 4.After menarche, before menopause.

Exclusion Criteria:

* 1. hormone therapy in the past 6 months. 2. Pregnancy in the past 6 months 3.Acute illness found in the past 3 months. 4.Systemic disease including autoimmune disease, malignancy, hepatic, renal or CVS disease, and ever received chemotherapy or immunosuppressive agents.

Ages: 17 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Dates: Start 2004-10; Study Completion 2005-08

CONTACTS AND LOCATIONS:
Overall Officials: Horng-Nerng Ho, M.D., Study Director — NTUH
Locations (1):
- Department of Obstetrics and Gynecology, National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Yang PK, Chou CH, Chang CH, Chen SU, Ho HN, Chen MJ. Changes in peripheral mitochondrial DNA copy number in metformin-treated women with polycystic ovary syndrome: a longitudinal study. Reprod Biol Endocrinol. 2020 Jul 13;18(1):69. doi: 10.1186/s12958-020-00629-5. PMID 32660613
- [Derived] Yang PK, Hsu CY, Chen MJ, Lai MY, Li ZR, Chen CH, Chen SU, Ho HN. The Efficacy of 24-Month Metformin for Improving Menses, Hormones, and Metabolic Profiles in Polycystic Ovary Syndrome. J Clin Endocrinol Metab. 2018 Mar 1;103(3):890-899. doi: 10.1210/jc.2017-01739. PMID 29325133